CLINICAL TRIAL: NCT06477744
Title: Long Term Follow-up of Patients With Parkinson's Disease Who Had Administered of Allogenic Embryonic Stem Cell-derived A9 Dopamine Progenitor Cell (A9-DPC) in SB-PD-001 Study
Brief Title: Long Term Follow-up of Patients With Parkinson's Disease Who Had Administered of A9-DPC in SB-PD-001 Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.Biomedics Co., Ltd. (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-PD-002
Record Dates: First submitted 2024-06-12; First posted 2024-06-27 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Group (Experimental): 1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Study group : 6 subjects
  3. Dosage: 3.15X10^6 cells/body (6 tracks in total, 52.5X10^4 cells per track)
  Interventions: Biological: Allogenic embryonic stem cellderived A9 dopamine progenitor cell (A9-DPC)_Low Dose
- High Dose Group (Experimental): 1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Study group : 6 subjects
  3. Dosage: 6.30X10^6 cells/body (6 tracks in total, 105X10^4 cells per track)
  Interventions: Biological: Allogenic embryonic stem cellderived A9 dopamine progenitor cell (A9-DPC)_High Dose

INTERVENTIONS:
Biological: Allogenic embryonic stem cellderived A9 dopamine progenitor cell (A9-DPC)_Low Dose — 1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Main ingredients and quantities: A9-DPC
     -Low Dose : 7.0X10^6 cells (Use 3.15X10^6 cells of this)
  3. Formulation: milky white cell suspension
  4. Storage method: Refrigerated storage (5±3℃)
  5. Expiration date: within 36 hours of manufacture
  6. Frequency: single dosing
  7. Method: The subject pierces a burr hole in the skull on the day of surgery. Then the cells are injected at a predetermined stem cell administration point of the putamen in the brain of the subject. One side is administered in three tracks per putamen (6 tracks total brain). Do the same for the other side.
  Arms: Low Dose Group
Biological: Allogenic embryonic stem cellderived A9 dopamine progenitor cell (A9-DPC)_High Dose — 1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Main ingredients and quantities: A9-DPC
     -High Dose : 1.4X10^7 cells (Use 6.30X10^6 cells of this)
  3. Formulation: milky white cell suspension
  4. Storage method: Refrigerated storage (5±3℃)
  5. Expiration date: within 36 hours of manufacture
  6. Frequency: single dosing
  7. Method: The subject pierces a burr hole in the skull on the day of surgery. Then the cells are injected at a predetermined stem cell administration point of the putamen in the brain of the subject. One side is administered in three tracks per putamen (6 tracks total brain). Do the same for the other side.
  Arms: High Dose Group

SUMMARY:
1. Long-term follow-up period: Approximately 72 months from the date of approval by the Institutional Review Board (IRB)( Study Period: From the A9-DPC treatment date of the first subject in SB-PD-001 Study* up to 5 years after the A9-DPC treatment of the last subject )
2. Objectives: This study aims to evaluate the long-term safety of A9-DPC by following up on the occurrence of adverse event of special interest, (AESI)* for 5 years from A9-DPC treatment date in subjects who have participated in SB-PD-001 Study and received A9-DPC. In addition, it will determine motor and non-motor symptoms over time following A9-DPC treatment, as measured by MDS-UPDRS.
3. Methods of the Long-term Follow-up : This is a single center, open-label, 5-year long-term follow-up to evaluate the long-term safety in subjects receiving A9-DPC in SB-PD-001 Study.

Among subjects who have received A9-DPC, those who have provided voluntary written informed consent for participation of the long-term follow-up will be included. The occurrence of AESIs is investigated for 5 years from A9-DPC treatment, and MDS-UPDRS will be conducted for the efficacy assessment if the study can be conducted.

To avoid any missing data about AESIs, a phone or site visit will be performed at least once yearly from the start of the follow-up.

DETAILED DESCRIPTION:
1. Population of the Long-term Follow-up : Subjects who have participated in SB-PD-001 Study and received A9-DPC (about 12 subjects)
2. Long-term Follow-up Period ; Approximately 72 months from the date of approval by the Institutional Review Board (IRB)

   * Study Period: From the A9-DPC treatment date of the first subject in SB-PD-001 Study* up to 5 years after the A9-DPC treatment of the last subject
   * Study Duration for Individual Subject: 5 years from A9-DPC treatment date * SB-PD-001 Study: Phase 1/2a study of A9-DPC
3. Objectives and Endpoints of the Long-term Follow-up ; This study aims to evaluate the long-term safety of A9-DPC by following up on the occurrence of adverse event of special interest, (AESI)* for 5 years from A9-DPC treatment date in subjects who have participated in SB-PD-001 Study and received A9-DPC. In addition, it will determine motor and non-motor symptoms over time following A9-DPC treatment, as measured by MDS-UPDRS.

   * AESI is a minimum investigation item to be observed for long-term follow-up of stem cell treatment among the adverse events (AEs) that occur in the subjects receiving treatment. In accordance with the Guideline for Long-term Follow-up of Advanced Biopharmaceuticals distributed by the Ministry of Food and Drug Safety in 2020, it is designated as below in this long-term follow-up. AESIs refer to the serious adverse events (SAEs) in the guideline.

   Adverse Event of Special Interests (AESIs)

   [Early-onset AESIs (up to 2 years* after the study drug treatment)]
   * Infectious diseases
   * Complications related to the associated surgical procedures

   [Late-onset AESIs (up to 5 years after the study drug treatment)]
   * Death
   * Generation of a neoplasm or malignant tumor in tissues or organs
   * Onset of an immune reaction including worsening of a previous autoimmune disease or new occurrence
   * Other delayed AESIs related to the treatment of embryonic stem cell-derived therapeutics.

   There is no delayed AESIs confirmed so far, and when any additional AESIs are detected in the subsequent follow-up, they will be added.
4. Drug under Long-term Follow-up ; Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
5. Inclusion Criteria ;

   * Persons who have participated in SB-PD-001 Study and received A9-DPC
   * Persons who have provided written informed consent for this long-term follow-up
6. Methods of the Long-term Follow-up ; This is a single center, open-label, 5-year long-term follow-up to evaluate the long-term safety in subjects receiving A9-DPC in SB-PD-001 Study.

   Among subjects who have received A9-DPC, those who have provided voluntary written informed consent for participation of the long-term follow-up will be included. The occurrence of AESIs is investigated for 5 years from A9-DPC treatment, and MDS-UPDRS will be conducted for the efficacy assessment if the study can be conducted.

   To avoid any missing data about AESIs, a phone or site visit will be performed at least once yearly from the start of the follow-up.
7. Analysis Methods ; Adverse Event of Special Interests (AESIs) For AESIs, the number of subjects affected, incidence rate, its exact 95% confidence interval (CI), and the number of events will be provided. In addition, the events will be coded using the Medical Dictionary For Regulatory Activities (MedDRA) with System Organ Class (SOC) and Preferred Term (PT), and the number of subjects affected, incidence rate, and the number of events will be provided.

MDS-UPDRS Total Score(defined On/Off), part Ⅲ (defined on/off) and IV score For changes at each time point after the IP treatment from baseline, descriptive statistics (number of subjects, mean, standard deviation, median, minimum, and maximum) will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have participated in SB-PD-001 Study and received A9-DPC.
* Persons who have provided written informed consent for this long-term follow-up.

Exclusion Criteria:

* Not Applicable

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2029-02-07 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Adverse Event of Special Interests (AESIs) | 5 years after IP administration
  Review occurrence of adverse event of special interests (AESIs)

SECONDARY OUTCOMES:
MDS-UPDRS Total Score (defined On/Off) | -Day 14 to -Day 4, 5 years after IP administration
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the MDS-UPDRS Total Scores, up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 14 to -Day 4).
  * Defined-on condition: condition that the most positive functional effect, as agreed by the subject and the tester, after treatment with drugs for controlling the symptoms of Parkinson's disease
  * Defined-off condition: condition after 12 hours off drugs for controlling the symptoms of Parkinson's disease
MDS-UPDRS part Ⅲ (defined On/Off) | -Day 14 to -Day 4, 5 years after IP administration
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the MDS-UPDRS part Ⅲ (defined On/Off) up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 14 to -Day 4).
  * Defined-on condition: condition that the most positive functional effect, as agreed by the subject and the tester, after treatment with drugs for controlling the symptoms of Parkinson's disease
  * Defined-off condition: condition after 12 hours off drugs for controlling the symptoms of Parkinson's disease
MDS-UPDRS Ⅳ score | -Day 14 to -Day 4, 5 years after IP administration
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the MDS-UPDRS Ⅳ score up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 14 to -Day 4).
  * Defined-on condition: condition that the most positive functional effect, as agreed by the subject and the tester, after treatment with drugs for controlling the symptoms of Parkinson's disease
  * Defined-off condition: condition after 12 hours off drugs for controlling the symptoms of Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Phil-hyu Lee, M.D.,Ph.D, Principal Investigator — Yonsei Universitiy Health System, Severance Hospital
Locations (1):
- Yonsei Universitiy Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendez I, Sanchez-Pernaute R, Cooper O, Vinuela A, Ferrari D, Bjorklund L, Dagher A, Isacson O. Cell type analysis of functional fetal dopamine cell suspension transplants in the striatum and substantia nigra of patients with Parkinson's disease. Brain. 2005 Jul;128(Pt 7):1498-510. doi: 10.1093/brain/awh510. Epub 2005 May 4. PMID 15872020
- [Background] Schweitzer JS, Song B, Herrington TM, Park TY, Lee N, Ko S, Jeon J, Cha Y, Kim K, Li Q, Henchcliffe C, Kaplitt M, Neff C, Rapalino O, Seo H, Lee IH, Kim J, Kim T, Petsko GA, Ritz J, Cohen BM, Kong SW, Leblanc P, Carter BS, Kim KS. Personalized iPSC-Derived Dopamine Progenitor Cells for Parkinson's Disease. N Engl J Med. 2020 May 14;382(20):1926-1932. doi: 10.1056/NEJMoa1915872. PMID 32402162
- [Background] Yasuhara T, Kameda M, Sasaki T, Tajiri N, Date I. Cell Therapy for Parkinson's Disease. Cell Transplant. 2017 Sep;26(9):1551-1559. doi: 10.1177/0963689717735411. PMID 29113472
- [Background] Kikuchi T, Morizane A, Doi D, Magotani H, Onoe H, Hayashi T, Mizuma H, Takara S, Takahashi R, Inoue H, Morita S, Yamamoto M, Okita K, Nakagawa M, Parmar M, Takahashi J. Human iPS cell-derived dopaminergic neurons function in a primate Parkinson's disease model. Nature. 2017 Aug 30;548(7669):592-596. doi: 10.1038/nature23664. PMID 28858313
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] National Institute of Food and Drug Safety, Ministry of Food and Drug Safety, Guideline for Long-term Follow-up of Advanced Biopharmaceuticals 2020.12
- [Background] Korea National Institute for Bioethics Policy, Instruction for Protection of Vulnerable Subjects 2019.7
- [Background] MDS-UPDRS Korean Official Translation. Last updated May 18, 2020.
- [Background] NCI-CTCAE v5.0 [Common Terminology Criteria for Adverse Events (CTCAE) (cancer.gov)]